CLINICAL TRIAL: NCT01347268
Title: A Prospective Randomized Study Comparing Coasting by Withholding GnRH Agonist With GnRH Antagonist Administration in Patients at Risk for Severe OHSS
Brief Title: Comparing Coasting by Withholding GnRH Agonist With GnRH Antagonist
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Jiann-Loung Hwang, Shin-Kong Wu Ho-Su Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SKH-8302-100-DR-08
Record Dates: First submitted 2011-04-26; First posted 2011-05-04 (Estimated); Last update posted 2011-05-04 (Estimated); Status verified 2011-01

CONDITIONS: In Vitro Fertilization
Keywords: coasting; withdrawing GnRH agonist; GnRH antagonist; IVF
MeSH Terms: interventions — LHRH, Ac-Nal(1)-Cpa(2)-Trp(3)-Arg(6)-Ala(10)-

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- withdrawing GnRH agonists (Experimental)
  Interventions: Procedure: withdrawing GnRH agonists
- GnRH antagonist administration (Experimental)
  Interventions: Procedure: GnRH antagonist

INTERVENTIONS:
Procedure: GnRH antagonist — GnRH antagonist administration and continued low dose r-FSH 75 IU
  Arms: GnRH antagonist administration
Procedure: withdrawing GnRH agonists — withdrawing GnRH agonists and continued low dose r-FSH 75 IU
  Arms: withdrawing GnRH agonists

SUMMARY:
Ovarian hyperstimulation syndrome (OHSS) is the most serious complication of ovulation induction and is a life threatening iatrogenic complication. In patients with GnRH agonist protocol, both withdrawing GnRH agonist and GnRH antagonist administration are associated with a reduction in (E2) levels with subsequent decreasing the incidence and severity of OHSS. This work is to compare the clinical and endocrine outcome response of cycles in which GnRH agonist withdrawing with cycles in which the GnRH antagonist administration in patients at risk of severe OHSS.

DETAILED DESCRIPTION:
Background: Elevated estradiol (E2) levels and multiple folliculogenesis predispose to development of ovarian hyperstimulation syndrome (OHSS). In patients with GnRH agonist protocol, both withdrawing GnRH agonist and GnRH antagonist administration are associated with a reduction in (E2) levels with subsequent decreasing the incidence and severity of OHSS. This work is to compare the clinical and endocrine outcome response of cycles in which GnRH agonist withdrawing with cycles in which the GnRH antagonist administration in patients at risk of severe OHSS.

Purpose: To compare the decreased levels of estradiol (E2), coasting days, severity of OHSS and pregnancy outcomes of cycles in which GnRH agonist withdrawing with cycles in which the GnRH antagonist administration in patients at risk of severe OHSS.

Methods: a prospective randomized study was designed to evaluate clinical and endocrine outcome in two different coasting protocols. Women (n=120) under controlled ovarian hyperstimulation with GnRH agonist protocol at the risk of OHSS (≧20 follicles >12 mm development with E2> 4000 pg/ml) randomized into two groups. Group I (n=60), withdrawing GnRH agonists and continued low dose r-FSH 75 IU. Group II (n=60), GnRH antagonist administration and continued low dose r-FSH 75 IU. When E2< 3000 pg/ml, hCG was given. Oocyte retrieval was performed 36 h after hCG administration. The primary outcome measures were the decreased levels of estradiol (E2) and the days of coasting. The secondary outcome measures were number of oocytes retrieved, pregnancy rate and the incidence of OHSS.

anticipated results: No significant differences were seen in the levels of estradiol (E2) decreased, the days of coasting, number of oocytes, pregnancy rate and the incidence of OHSS. GnRH antagonist is not necessary in coasting treatment while stop GnRH agonist.

ELIGIBILITY:
Inclusion Criteria:

* the risk of ovarian hyperstimulation syndrome

Exclusion Criteria:

* allergic to GnRH antagonist

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-06 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
decreased levels of estradiol (E2) | one year
The days of coasting | one year
  The interval between the day of starting intervention and the day of hCG administration

SECONDARY OUTCOMES:
number of oocytes retrieved | one year
pregnancy rate | one year
the incidencess of OHSS | one year

CONTACTS AND LOCATIONS:
Overall Officials: Jiann-Loung Hwang, MD, Study Chair — Shin-Kong Wu Ho-Su Memerial Hospital
Locations (1):
- Department of Obstetrics and Gynecology, Shin-Kong Wu Ho-Su Memerial Hospital, Taipei, Taiwan